CLINICAL TRIAL: NCT00543257
Title: Parents at the Center: Information Management in ADHD - Clinical Trial
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Eugenia Chan, Assistant In Medicine, Boston Children's Hospital
Other Study IDs: CHB-R01LM009256
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Health Literacy; Attention Deficit Disorder With Hyperactivity; Computer Literacy; Information Management; Parents
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parents: Parents of children with ADHD will be recruited from the greater Boston community. We are interested in enrollment of parents with a range of educational and technical backgrounds, and specifically will look to enroll parents who may not have much computer experience.
  Interventions: Other: Use of paper forms to write down information; Other: Computer

INTERVENTIONS:
Other: Use of paper forms to write down information — Parents will be asked to write down information specific to their child's ADHD using paper forms.
Other: Computer — Parents will use a computer to complete data entry on information specific to their child's ADHD care

SUMMARY:
Health literacy is an integral part of the pathway for the successful transfer of information between patients and providers. Parents of children with Attention Deficit/ Hyperactivity Disorder (ADHD) play an essential role in chronic care as they offer critical information to providers that drives appropriate education and disease management. We propose the development and evaluation of an electronic data entry tool that enables parents to communicate data essential to treatment of their children, regardless of their own literacy skills. The research plan addresses a question central to patient-centered information management: how does health literacy influence parents' report of data on ADHD and the process-level events that result from parent-provider communication? The following specific aims organize the clinical study: proposal: 1) To assess the effect of health literacy on successful completion of parent-reported ADHD health information in both paper-based and PCHR formats, and, 2): To determine the association between health literacy and process-level outcomes for ADHD that stem from parent-provider exchange of information. The formal evaluation will study a diverse cohort of parents in a randomized trial of data entry (paper versus PCHR) for ADHD-specific information. Primary care records for children of this cohort will be analyzed for the prior 12 month period. Both a retrospective examination of documented ADHD processes of care and a prospective evaluation of the utility of data from the PCHR will occur. Literacy level is a primary variable of interest throughout the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Primary language of parent/guardian is English or Spanish
* Parent/guardian reports that child has been diagnosed with ADHD
* Current child age is between 5 years and 12 years
* Child in question resides with the parental subject primarily
* Parent/guardian reports that they are the primary caretaker of the child
* Parent/guardian reports that they are the person who communicates with the primary care provider
* Parent/guardian reports that child is currently taking medication for ADHD or has taken it within the last 3 months

Exclusion Criteria:

* Parent reports that child in question has been diagnosed with mental retardation, autism, pervasive developmental disorder, Aspergers, or bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents of school-age children with ADHD
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Porter, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Porter SC, Guo CY, Bacic J, Chan E. Health literacy and task environment influence parents' burden for data entry on child-specific health information: randomized controlled trial. J Med Internet Res. 2011 Jan 26;13(1):e13. doi: 10.2196/jmir.1612. PMID 21269990